CLINICAL TRIAL: NCT02606084
Title: An Open-Label, Single-Dose, Parallel-Group Study to Assess the Effects of Renal Impairment on the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine
Brief Title: A Study to Assess the Effects of Renal Impairment on the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108058; 54135419TRD1014 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Renal Impairment; Healthy
Keywords: Renal Impairment; Healthy; Esketamine
MeSH Terms: conditions — Renal Insufficiency | interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants with mild renal impairment (Measured Creatinine Clearance [CLCR,m] greater than or equal to >= 50 to 79 milliliter/minute [mL/min]) will self-administer esketamine 28 milligram (mg) intranasally on Day 1.
  Interventions: Drug: Esketamine
- Cohort 2 (Experimental): Participants with moderate renal impairment (CLCR,m >=30 to 49 mL/min) will self-administer esketamine 28 mg intranasally on Day 1.
  Interventions: Drug: Esketamine
- Cohort 3 (Experimental): Participants with severe renal impairment (CLCR,m less than [<] 30 mL/min), not on dialysis will self-administer esketamine 28 mg intranasally on Day 1.
  Interventions: Drug: Esketamine
- Cohort 4 (Experimental): Participants with normal renal function and no evidence of kidney damage (CLCR,m >= 80 mL/min) will self-administer esketamine 28 mg intranasally on Day 1.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — Participants will self-administer esketamine solution intranasally 28 milligram (mg) on Day 1.
  Other Names: JNJ-54135419

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of a single dose of intranasally administered esketamine in participants with impaired renal function when compared to participants with normal renal function.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-dose, single-center, parallel group study to characterize the pharmacokinetics and safety of a single 28 milligram (mg) dose of esketamine in both participants with varying stages of renal impairment and healthy participants. A total of approximately 32 medically stable men and women with varying degrees of renal function impairment or no renal impairment will be enrolled. The study consists of a Screening period of up to Days -21 to -2, open label phase of Days -1 to 4, and end-of-study (11 plus [+] or minus [-] 2 days after final dose). The participants will be assigned to 1 of 4 groups (8 participants per group) based on creatinine clearance (CLCR,m). Safety and tolerability will be assessed from the time of consent until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* For women of childbearing potential, must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at Screening; and a negative urine pregnancy test on Day minus (-) 1
* Comfortable with self-administration of intranasal medication and able to follow instructions provided
* Hemoglobin concentration of greater than or equal to (>=) 10 grams per deciLiter (g/dL) (Only for cohorts 1, 2, and 3)
* Platelet count of >= 50,000 counts/microliter (Only for cohorts 1, 2, and 3)

Exclusion Criteria:

* Current or previous diagnosis of psychotic or major depressive disorder (MDD) with psychosis, bipolar or related disorder, intellectual disability, borderline personality disorder, or antisocial personality disorder
* A lifetime history of cerebrovascular disease including stroke or transient ischemic attack, aneurysmal vascular disease
* Unstable coronary artery disease or myocardial infarction in the last 12 months or any unstable angina requiring revascularization procedure, hemodynamically significant valvular heart disease, or New York Heart Association Class III-IV heart failure
* Has had a renal transplant or diagnosis of systemic lupus erythromatosus or renal carcinoma
* Has a nasal piercing
* Participant requires dialysis (Only for cohorts 1, 2, and 3)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 60 hours post-dose
  The Cmax is the maximum observed concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 60 hours post-dose
  The Tmax is defined as actual sampling time to reach maximum observed concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | 60 hours post-dose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | 60 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C(last)/lambda(z); wherein AUC (last) is area under the plasma concentration time curve from time zero to last quantifiable time, C (last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Elimination Rate Constant (Lambda[z]) | 60 hours post-dose
  Lambda (z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Amount of Drug excreted in Urine (Ae) | 60 hours post-dose
  Total amount excreted into the urine, calculated as the sum of all Ae(t1-t2) intervals.
Measured Creatinine Clearance (CLCR,m) | 60 hours post-dose
Estimated Creatinine Clearance (CLCR,e) | 60 hours post-dose

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Screening up to End of Follow-up Phase (approximately up to 34 - 38 days)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Miami, Florida
  - Knoxville, Tennessee

REFERENCES:
- See also: An Open-Label, Single-Dose, Parallel-Group Study to Assess the Effects of Renal Impairment on the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108058&attachmentIdentifier=f5911918-6048-4dec-8e77-5fc22104b6ae&fileName=CR108058_CSR.pdf&versionIdentifier=